CLINICAL TRIAL: NCT01967173
Title: Best African American Response to Asthma Drugs
Acronym: BARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 006; 1U10HL098115 (NIH)
Record Dates: First submitted 2013-10-11; First posted 2013-10-22 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone; Salmeterol
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Crossover sequence 1 (Experimental): Flovent Diskus® 250 mcg,followed by Advair Diskus® 250/50 mcg, followed by Flovent Diskus® 100 mcg, followed by Advair Diskus® 100/50 mcg
  Interventions: Drug: Flovent Diskus® 100 mcg; Drug: Flovent Diskus® 250 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 2 (Experimental): Advair Diskus® 250/50 mcg, followed by Advair Diskus® 100/50 mcg, followed by Flovent Diskus® 250 mcg, followed by Flovent Diskus® 100 mcg
  Interventions: Drug: Flovent Diskus® 100 mcg; Drug: Flovent Diskus® 250 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 3 (Experimental): Flovent Diskus® 100 mcg, followed by Flovent Diskus® 250 mcg, followed by Advair Diskus® 100/50 mcg, followed by Advair Diskus® 250/50 mcg
  Interventions: Drug: Flovent Diskus® 100 mcg; Drug: Flovent Diskus® 250 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 4 (Experimental): Advair Diskus® 100/50 mcg, followed by Flovent Diskus® 100 mcg, followed by Advair Diskus® 250/50 mcg, followed by Flovent Diskus® 250 mcg
  Interventions: Drug: Flovent Diskus® 100 mcg; Drug: Flovent Diskus® 250 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 5 (Experimental): Flovent Diskus® 500 mcg, followed by Advair Diskus® 250/50 mcg, followed by Flovent Diskus® 250 mcg, followed by Advair Diskus® 100/50 mcg
  Interventions: Drug: Flovent Diskus® 250 mcg; Drug: Flovent Diskus® 500 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 6 (Experimental): Advair Diskus® 250/50 mcg, followed by Advair Diskus® 100/50 mcg, followed by Flovent Diskus® 500 mcg, followed by Flovent Diskus® 250 mcg
  Interventions: Drug: Flovent Diskus® 250 mcg; Drug: Flovent Diskus® 500 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 7 (Experimental): Flovent Diskus® 250 mcg, followed by Flovent Diskus® 500 mcg, followed by Advair Diskus® 100/50 mcg, followed by Advair Diskus® 250/50 mcg
  Interventions: Drug: Flovent Diskus® 250 mcg; Drug: Flovent Diskus® 500 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg
- Crossover sequence 8 (Experimental): Advair Diskus® 100/50 mcg, followed by Flovent Diskus® 250 mcg, followed by Advair Diskus® 250/50 mcg, followed by Flovent Diskus® 500 mcg
  Interventions: Drug: Flovent Diskus® 250 mcg; Drug: Flovent Diskus® 500 mcg; Drug: Advair Diskus® 100/50 mcg; Drug: Advair Diskus® 250/50 mcg

INTERVENTIONS:
Drug: Flovent Diskus® 100 mcg — Flovent is an ICS
  Arms: Crossover sequence 1; Crossover sequence 2; Crossover sequence 3; Crossover sequence 4
Drug: Flovent Diskus® 250 mcg — Flovent is an ICS
Drug: Flovent Diskus® 500 mcg — Flovent is an ICS
  Arms: Crossover sequence 5; Crossover sequence 6; Crossover sequence 7; Crossover sequence 8
Drug: Advair Diskus® 100/50 mcg — Advair is an ICS/LABA combination
Drug: Advair Diskus® 250/50 mcg — Advair is an ICS/LABA combination

SUMMARY:
The purpose of this study is to find the best asthma treatment to add for Blacks who have asthma that is not well controlled on a low dose of inhaled steroid. This study will also try to find out if Black adults and children differ in how they respond to the medications used in this study.

DETAILED DESCRIPTION:
BARD is a 66 week prospective, randomized, double-blind, crossover trial in Blacks (individuals who self-report Black ancestry) who have inadequately controlled asthma while taking low-dose inhaled corticosteroids (ICS). BARD will examine the efficacy of increasing the dose of ICS with or without the addition of a long-acting beta agonist (LABA) to determine whether individual patients respond better to one treatment than another and, if so, whether the responses are different for children and adults or if they are related to genetic ancestry.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who self-report Black ancestry (with at least 1 Black grandparent).
2. Able to perform reproducible spirometry according to ATS criteria.
3. Clinical history consistent with asthma.
4. Baseline FEV1≥40% of predicted and/or post-bronchodilator FEV1≥40% of predicted.
5. Asthma confirmed either by: (1) Beta-agonist reversibility to 4 puffs albuterol ≥ 12% OR (2) PC20FEV1 ≤ 16 mg/ml OR (3) an absolute relative change in %predicted FEV1 of ≥ 12% over two measurements documented by repeat spirogram over the previous year
6. Either: A) inadequately controlled on low-, medium- or high-dose ICS monotherapy, or low- or medium-dose ICS/LABA, or B) well-controlled on medium- or high-dose ICS monotherapy, or low-, medium- or high-dose ICS/LABA. Inadequate asthma control will be defined as an ACT/c-ACT score <20; well-controlled asthma will be defined as an ACT/c-ACT score ≥20.
7. Stable asthma controller therapy dose (ICS or ICS/LABA) for the 2 weeks prior to enrollment.
8. Non-smoker (total lifetime smoking history < 5 pack-years if <18, or <10 pack-years if ≥18 years of age; no smoking for at least 1 year).
9. For participants ≥18 years of age: Ability to provide informed consent. For participants under 18 years of age: Ability to provide verbal or written assent and ability of parent to provide informed consent.

Exclusion Criteria:

1. Medical contraindication to LABA or history of adverse reactions to ICS or LABA preparations or any of their ingredients.
2. Current or prior use of medications known to significantly interact with corticosteroid disposition within the two-week period preceding enrollment.
3. Unwilling to provide a blood sample for DNA extraction and genetic analysis.
4. Major medical problems prohibiting study participation, i.e. presence of chronic or active lung disease other than asthma or history of unstable significant medical illness other than asthma, including thyroid disease, diabetes mellitus, Cushing's disease, Addison's disease, hepatic disease, or concurrent medical problems that could require oral corticosteroids during the study or that would place the participant at increased risk.
5. Systemic corticosteroid treatment for any condition within 4 weeks of enrollment or more than five courses of systemic corticosteroids in the past year.
6. History of a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure within the last 2 years.
7. History of a respiratory tract infection within 4 weeks of enrollment.
8. If a female of child-bearing potential, failure to practice abstinence or use an acceptable birth control method.
9. Pregnancy or lactation or planning to get pregnant during the course of the trial.
10. Receiving hyposensitization therapy other than an established maintenance regimen defined as a continuous regimen for ≥ 3 months prior to enrollment.
11. Participation in an intervention trial or use of investigative drugs in the past 30 days or plans to enroll in such a trial during the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2014-02; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (28):
- United States (28):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of California - San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Case Western Reserve University, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Center for Urban Population Health, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Wechsler ME, Szefler SJ, Ortega VE, Pongracic JA, Chinchilli V, Lima JJ, Krishnan JA, Kunselman SJ, Mauger D, Bleecker ER, Bacharier LB, Beigelman A, Benson M, Blake KV, Cabana MD, Cardet JC, Castro M, Chmiel JF, Covar R, Denlinger L, DiMango E, Fitzpatrick AM, Gentile D, Grossman N, Holguin F, Jackson DJ, Kumar H, Kraft M, LaForce CF, Lang J, Lazarus SC, Lemanske RF Jr, Long D, Lugogo N, Martinez F, Meyers DA, Moore WC, Moy J, Naureckas E, Olin JT, Peters SP, Phipatanakul W, Que L, Raissy H, Robison RG, Ross K, Sheehan W, Smith LJ, Solway J, Sorkness CA, Sullivan-Vedder L, Wenzel S, White S, Israel E; NHLBI AsthmaNet. Step-Up Therapy in Black Children and Adults with Poorly Controlled Asthma. N Engl J Med. 2019 Sep 26;381(13):1227-1239. doi: 10.1056/NEJMoa1905560. PMID 31553835
- See also: AsthmaNet — http://asthmanetresearch.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6 | Crossover Sequence 7 | Crossover Sequence 8
Started | 69 | 69 | 71 | 71 | 73 | 72 | 75 | 74
Completed 1st Period | 58 | 60 | 67 | 65 | 64 | 62 | 67 | 69
Completed 2nd Period | 52 | 58 | 63 | 62 | 63 | 57 | 63 | 61
Completed 3rd Period | 48 | 54 | 60 | 61 | 59 | 56 | 59 | 56
Completed 4th Period | 45 | 52 | 55 | 57 | 56 | 49 | 57 | 50
Completed | 45 | 52 | 55 | 57 | 56 | 49 | 57 | 50
Not Completed | 24 | 17 | 16 | 14 | 17 | 23 | 18 | 24
Not completed — Lost to Follow-up | 5 | 3 | 2 | 4 | 8 | 12 | 6 | 8
Not completed — Physician Decision | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 14 | 10 | 7 | 8 | 9 | 10 | 12

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6 | Crossover Sequence 7 | Crossover Sequence 8 | Total
Number analyzed (Participants) | 69 | 69 | 71 | 71 | 73 | 72 | 75 | 74 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (2.0) | 8.5 (1.7) | 8.4 (1.9) | 8.4 (1.8) | 38.5 (16.5) | 38.5 (15.9) | 39.3 (16.0) | 35.6 (16.0) | 23.2 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 26 | 28 | 52 | 48 | 47 | 52 | 309
  Male | 40 | 42 | 45 | 43 | 21 | 24 | 28 | 22 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 7 | 6 | 2 | 2 | 2 | 3 | 33
  Not Hispanic or Latino | 62 | 65 | 64 | 65 | 71 | 70 | 73 | 71 | 541
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 63 | 65 | 68 | 66 | 69 | 71 | 74 | 73 | 549
  Other | 6 | 4 | 3 | 5 | 4 | 1 | 1 | 1 | 25
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 71 | 71 | 73 | 72 | 75 | 74 | 574
Forced expiratory volume at one second (FEV1) Percent of Predicted [Mean (Standard Deviation); unit: percent] — FEV1, expressed as percent of predicted FEV1 based on age, sex, race, and height.
  percent | 98.1 (15.4) | 92.6 (17.9) | 95 (13.6) | 96.2 (19.1) | 83.8 (19.1) | 82.9 (15.5) | 83.7 (17.3) | 83.4 (18) | 89.3 (18.1)
Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — Asthma Control Test: The score is calculated as the sum total of a 5-item questionnaire. Each item ranges from 1 (poor control) to 5 (good control) so that the range of the total score is 5 to 25. Scores below 20 indicate that asthma is not well controlled. Population: Asthma Control Test is not validated for use in children
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 73 | 72 | 75 | 74 | 294
    (all) |  |  |  |  | 18.9 (3.8) | 18.6 (3.9) | 19.2 (3.7) | 18.8 (3.8) | 18.9 (3.8)
Childhood Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — Childhood Asthma Control Test is for children 4-11 years of age: The score is calculated as the sum total of a 7-item questionnaire. Four items ranges from 0 (poor control) to 3 (good control) and three items ranges from 0 (poor control) to 5 (good control) so so that the range of the total score is 0 to 27. Scores below 20 indicate that asthma is not well controlled. Population: Childhood Asthma Control Test is not validated for use in adults
  units on a scale
    number analyzed (Participants) | 69 | 69 | 71 | 71 | 0 | 0 | 0 | 0 | 280
    (all) | 21.5 (3.7) | 21.2 (3.6) | 20.7 (4.1) | 22.1 (3.6) |  |  |  |  | 21.4 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is a Composite Measure That Uses Exacerbations, Asthma Control Days During the Last 12 of 14 Weeks of a Treatment Regimen, and Percent Predicted FEV1 at the End of a Treatment Regimen.
Description: This composite outcome uses a hierarchical method to ascertain differences in asthma control. For each participant, treatments are first compared to see if they differ in terms of exacerbations. If one treatment results in fewer exacerbations than another, it is deemed the superior treatment and no further comparisons are made. If treatment superiority cannot be assigned by exacerbations, then they are compared by asthma control days (ACDs). If one treatment yields at least 31 annualized ACDs more than another, it is deemed the superior treatment. If treatment superiority still cannot be assigned by ACDs, then they are compared by percent predicted FEV1 at the end of a treatment period. If one treatment yields at least 5% greater FEV1 than another, it is deemed the superior treatment. If treatment superiority cannot be assigned by exacerbations, ACDs or FEV1, then that participant is classified as having no differential response.
Time Frame: The last 12 weeks of each 14-week treatment period
Population: Not all treatments were used in all participants. Flovent 500 was not used in children and Flovent 100 was not used in adolescents and adults
Measure: Number; unit: probability
Groups:
- Adolescents and Adults: All study participant age 12 years or greater
- Children: All study participants under age 12 years
Arm/Group | Adolescents and Adults | Children
Number analyzed (Participants) | 294 | 280
probability
  Advair 100/50 superior to Flovent 250 | .49 | .46
  Advair 100/50 inferior to Flovent 250 | .28 | .46
  Advair 100/50 superior to Flovent 500: number analyzed (Participants) | 294 | 0
  Advair 100/50 superior to Flovent 500 | .53 |
  Advair 100/50 inferior to Flovent 500: number analyzed (Participants) | 294 | 0
  Advair 100/50 inferior to Flovent 500 | .27 |
  Advair 100/50 superior to Advair 250/50 | .42 | .47
  Advair 100/50 inferior to Advair 250/50 | .36 | .49
  Advair 100/50 superior to Flovent 100: number analyzed (Participants) | 0 | 280
  Advair 100/50 superior to Flovent 100 |  | .53
  Advair 100/50 inferior to Flovent 100: number analyzed (Participants) | 0 | 280
  Advair 100/50 inferior to Flovent 100 |  | .41
  Advair 250/50 superior to Flovent 250 | .46 | .43
  Advair 250/50 inferior to Flovent 250 | .33 | .47
  Advair 250/50 superior to Flovent 500: number analyzed (Participants) | 294 | 0
  Advair 250/50 superior to Flovent 500 | .49 |
  Advair 250/50 inferior to Flovent 500: number analyzed (Participants) | 294 | 0
  Advair 250/50 inferior to Flovent 500 | .31 |
  Flovent 500 superior to Flovent 250: number analyzed (Participants) | 294 | 0
  Flovent 500 superior to Flovent 250 | .35 |
  Flovent 500 inferior to Flovent 250: number analyzed (Participants) | 294 | 0
  Flovent 500 inferior to Flovent 250 | .40 |
  Flovent 250 superior to Flovent 100: number analyzed (Participants) | 0 | 280
  Flovent 250 superior to Flovent 100 |  | .51
  Flovent 250 inferior to Flovent 100: number analyzed (Participants) | 0 | 280
  Flovent 250 inferior to Flovent 100 |  | .37
Statistical Analysis 1: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Advair 100/50 compared to Fluticasone 250 is equal to the inferiority of Advair 100/50 compared to Fluticasone 250; Test type: Superiority; p = 0.003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Children; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9, Mixed Models Analysis
Statistical Analysis 3: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Advair 100/50 compared to Fluticasone 500 is equal to the inferiority of Advair 100/50 compared to Fluticasone 500; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Advair 100/50 compared to Advair 250/50 is equal to the inferiority of Advair 100/50 compared to Advair 250/50; Test type: Superiority; p = 0.42, Mixed Models Analysis
Statistical Analysis 5: Comparison: Children; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.84, Mixed Models Analysis
Statistical Analysis 6: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Advair 250/50 compared to Fluticasone 500 is equal to the inferiority of Advair 250/50 compared to Fluticasone 500; Test type: Superiority; p = 0.015, Mixed Models Analysis
Statistical Analysis 7: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Advair 250/50 compared to Fluticasone 250 is equal to the inferiority of Advair 250/50 compared to Fluticasone 250; Test type: Superiority; p = 0.085, Mixed Models Analysis
Statistical Analysis 8: Comparison: Children; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.62, Mixed Models Analysis
Statistical Analysis 9: Comparison: Adolescents and Adults; Test of the null hypothesis that the superiority of Fluticasone 500 compared to Fluticasone 250 is equal to the inferiority of Fluticasone 500 compared to Fluticasone 250; Test type: Superiority; p = 0.48, Mixed Models Analysis
Statistical Analysis 10: Comparison: Children; Test of the null hypothesis that the superiority of Advair 100/50 compared to Fluticasone 100 is equal to the inferiority of Advair 100/50 compared to Fluticasone 100; Test type: Superiority; p = 0.14, Mixed Models Analysis
Statistical Analysis 11: Comparison: Children; Test of the null hypothesis that the superiority of Fluticasone 250 compared to Fluticasone 100 is equal to the inferiority of Fluticasone 250 compared to Fluticasone 100; Test type: Superiority; p = 0.096, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Each participant was followed over the course of four 14-week treatment periods for a total of 56 weeks. The adverse events recorded below are reported at the treatment period level and represent 14 weeks of "at risk" exposure time.
Groups:
- Flovent 250 in Pediatric Group: Flovent 250 in participants under 12 years
- Advair 250/50 in Pediatric Group: Advair 250/50 in participants under 12 years
- Flovent 100 in Pediatric Group: Flovent 100 in participants under 12 years
- Advair 100/50 in Pediatric Group: Advair 100/50 in participants under 12 years
- Flovent 500 in Adolescent/Adult Group: Flovent 500 in participants 12 years and older
- Advair 250/50 in Adolescent/Adult Group: Advair 250/50 in participants 12 years and older
- Flovent 250 in Adolescent/Adult Group: Flovent 250 in participants 12 years and older
- Advair 100/50 in Adolescent/Adult Group: Advair 100/50 in participants 12 years and older
Arm/Group | Flovent 250 in Pediatric Group | Advair 250/50 in Pediatric Group | Flovent 100 in Pediatric Group | Advair 100/50 in Pediatric Group | Flovent 500 in Adolescent/Adult Group | Advair 250/50 in Adolescent/Adult Group | Flovent 250 in Adolescent/Adult Group | Advair 100/50 in Adolescent/Adult Group
All-Cause Mortality (participants affected / at risk) | 0/280 | 0/280 | 0/280 | 0/280 | 0/294 | 0/294 | 0/294 | 0/294
Serious Adverse Events (participants affected / at risk) | 8/280 | 1/280 | 2/280 | 4/280 | 10/294 | 7/294 | 7/294 | 8/294
Other Adverse Events (participants affected / at risk) | 64/280 | 52/280 | 43/280 | 27/280 | 53/294 | 47/294 | 35/294 | 34/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent 250 in Pediatric Group (N=280) | Advair 250/50 in Pediatric Group (N=280) | Flovent 100 in Pediatric Group (N=280) | Advair 100/50 in Pediatric Group (N=280) | Flovent 500 in Adolescent/Adult Group (N=294) | Advair 250/50 in Adolescent/Adult Group (N=294) | Flovent 250 in Adolescent/Adult Group (N=294) | Advair 100/50 in Adolescent/Adult Group (N=294)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Peptic Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar Spinal Cord Compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Post-Op Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse Food Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic Shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Closed Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug Withdrawal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intermittent Explosive Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Neoplasm Brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant Neoplasm Thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain Not Elsewhere Classified (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsions Not Elsewhere Classified (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope and Collapse (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent 250 in Pediatric Group (N=280) | Advair 250/50 in Pediatric Group (N=280) | Flovent 100 in Pediatric Group (N=280) | Advair 100/50 in Pediatric Group (N=280) | Flovent 500 in Adolescent/Adult Group (N=294) | Advair 250/50 in Adolescent/Adult Group (N=294) | Flovent 250 in Adolescent/Adult Group (N=294) | Advair 100/50 in Adolescent/Adult Group (N=294)
Acute Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 20 (35) | 18 (36) | 19 (33) | 20 (39) | 24 (33) | 27 (46) | 20 (40) | 22 (42)
Acute Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 16 (25) | 10 (14) | 11 (16) | 11 (20) | 11 (19) | 11 (15) | 16 (24) | 13 (20)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 23 (41) | 20 (47) | 40 (54) | 18 (31) | 18 (20) | 17 (20) | 17 (22) | 18 (23)
Cough (General disorders) | 11 (20) | 10 (23) | 13 (24) | 15 (21) | 2 (2) | 3 (5) | 6 (7) | 3 (3)
Fever (General disorders) | 10 (11) | 6 (8) | 16 (19) | 8 (10) | 4 (4) | 3 (3) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT01967173/Prot_SAP_000.pdf